CLINICAL TRIAL: NCT02417662
Title: Stereotactic Ablative Radiotherapy for Oligometastatic Non-small Cell Lung Cancer. a Randomised Phase III Trial
Brief Title: Stereotactic Ablative Radiotherapy for Oligometastatic Non-small Cell Lung Cancer
Acronym: SARON
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL/13/0594
Record Dates: First submitted 2015-03-20; First posted 2015-04-16 (Estimated); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; Stereotactic Ablative Radiotherapy; Radiotherapy; Randomised; Controlled; Oligometastatic
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Systemic Anti-Cancer Therapy (SACT) alone (Active Comparator): The choice of SACT is determined by the treating clinician and will be supplied from hospital commercial stock, and prepared and administered according to institutional guidelines.
  Interventions: Other: Non-investigational SACT
- SACT + Radical Radiotherapy (Conventional RT and SABR) (Experimental): SACT followed by radical RT (conventional or SABR) to the primary and SABR to the metastatic sites.
  The choice of SACT is determined by the treating clinician and will be supplied from hospital commercial stock, and prepared and administered according to institutional guidelines.
  Interventions: Radiation: Radical Radiotherapy (Conventional RT and SABR)

INTERVENTIONS:
Radiation: Radical Radiotherapy (Conventional RT and SABR) — Radical radiotherapy (conventional or SABR) to primary and SABR to the metastases
  Arms: SACT + Radical Radiotherapy (Conventional RT and SABR)
Other: Non-investigational SACT — There is no intervention in the control group, patients will receive SACT. The choice of SACT is determined by the treating clinician and will be supplied from hospital commercial stock, and prepared and administered according to institutional guidelines.
  Arms: Systemic Anti-Cancer Therapy (SACT) alone

SUMMARY:
The trial will assess the addition of stereotactic ablative radiotherapy (SABR) to standard anti-cancer therapy (SACT) in patients with oligometastatic non-small cell lung cancer. Patients will be randomised to receive either standard treatment alone (SACT) or standard treatment with conventional radiotherapy (RT) and SABR.

DETAILED DESCRIPTION:
SARON is a confirmatory phase III study examining the efficacy and safety of stereotactic ablative radiotherapy (SABR) and conventional radiotherapy (RT) alongside standard chemotherapy in patients with oligometastatic non-small cell lung cancer.

Current treatment for this group of patients is systemic anti-cancer therapy. The choice of SACT is determined by the treating clinician and will be supplied from hospital commercial stock, and prepared and administered according to institutional guidelines. There is sufficient evidence regarding the safety of SABR, its effect on local control and a possible impact on overall survival. This trial will further examine overall survival, progression free survival and local control, as well as toxicity, feasibility, patient reported outcomes and health resource use.

There will be a feasibility analysis performed after 50 patients have been randomised. This will assess the practicality of achieving recruitment targets, logistics of delivering the experimental treatment and the potential for contamination (as patients may seek SABR outside of the trial if randomised to the non SABR arm). There will also be a parallel thoracic SABR safety and feasibility study after recruitment and treatment of 20 patients with thoracic metastases.

This is a multicentre randomised phase III study based on patients with oligometastatic NSCLC.

Trial arms:

Control Arm: systemic anti-cancer therapy alone (SACT) Experimental Arm: SACT plus radical RT to primary and SABR and/or SRS to metastases

ELIGIBILITY:
Registration Inclusion criteria

1. Patient ≥ 18 years
2. Histologically or cytologically confirmed NSCLC.
3. Staging with FDG PET-CT whole body scan and MRI brain within 45 days prior to registration (but prior to commencement of first cycle of SACT). [Note: Brain CT with IV contrast can be performed instead (within 45 days prior to registration). However, if brain metastases are evident on the brain CT then a brain MRI must be performed prior to randomisation, i.e. the Brain CT is sufficient for registration into the trial but not for randomisation if it is positive for brain metastases, in which case a brain MRI must be performed]
4. ECOG performance status 0 to 1 (prior to commencement of first cycle of SACT).
5. Patient presenting with primary disease +/- lymph nodes and synchronous oligometastatic disease (1-5 lesions in up to a maximum of 3 organs).
6. Patient is deemed fit to receive four cycles of systemic anti-cancer therapy, according to local guidelines and assessment.
7. Patient is deemed fit to receive radical RT (either conventional RT or SABR) to primary disease +/- lymph node and SABR/SRS to 1-5 metastases according to local guidelines and assessment.
8. Primary tumour +/- lymph node suitable for radical RT (either conventional RT or SABR).
9. 1-5 metastatic lesions in up to a maximum of 3 organs, assessable according to RECIST v1.1 and all of which are suitable for SABR/SRS (only one site of metastasis or primary tumour needs to be measurable according to RECIST v1.1).

   i. If brain metastasis present, the NHS commissioning guidelines need to be met for intracranial SRS (≤20 cc) (or equivalent for Wales, Scotland & Northern Ireland in line with standard of care).

   ii. Lymph nodes included in the N1-3 categories of the IASLC 2009 staging criteria are treated in the conventional radiotherapy volume and are not counted as metastases.

   iii. Lymph nodes not included in the N1-3 categories of the IASLC 2009 staging criteria, e.g. pelvic lymph nodes, are counted as metastases.

   iv. For bone metastases pre-SABR stabilisation should be considered as clinically appropriate. This does not exclude the patient from the study.
10. Acceptable lung function for radical lung radiotherapy as assessed according to local policy. Note: Potential thoracic sub-study patients will need to complete pulmonary function tests pre-randomisation
11. No relevant co-morbidities, including UIP pulmonary fibrosis and connective tissue disorders.

Additional inclusion Information Patients with lung cancer and an additional malignant nodule are difficult to categorise, and the current stage classification rules are unclear. Such patients should be evaluated by the local multidisciplinary team to determine whether the additional lesion represents a second primary lung cancer or an additional tumour nodule corresponding to the dominant cancer. The SARON TMG will accept local MDM decisions on this and will centrally review all baseline imaging retrospectively

Registration Exclusion Criteria

1. Patient has had palliative radiotherapy to any tumour site prior to registration or requires palliative radiotherapy prior to randomisation.
2. Presence of an actionable molecular aberration.
3. Patients currently receiving VEGF inhibitors.
4. One or more metastases previously treated with alternative ablative treatment.Note: Surgical ablation (partial or total excision biopsy) is permitted for palliative or diagnostic purposes (e.g. for molecular analysis). Treatment for any residual disease/tumour bed will be at the discretion of treating clinician/MDT. Resected/ablated metastases will count towards the total number of metastases.
5. Patient has received any previous treatment for this NSCLC malignancy.
6. Patients who present with brain metastasis only and no sites of extra cranial metastatic disease i.e. the presence of more than 4 brain metastases is an exclusion criterion.
7. Metastasis in sites where normal radiotherapy OAR constraints cannot be met.
8. Brain metastasis within the brainstem.
9. Patients who have more than five sites of metastases in up to 3 organs prior to trial registration.
10. Primary tumour or metastases causing direct invasion or high clinical suspicion of direct invasion of the wall of a major blood vessel, oesophagus, trachea, proximal bronchial tree, stomach, intestines or mesenteric lymph nodes or cutaneous metastases or diffuse serosal metastases.
11. Malignant pleural or pericardial effusion.
12. Bilateral adrenal metastases.
13. History of prior malignant tumour likely to interfere with the protocol treatment, (patients without evidence of disease for at least 1 year or a non-melanoma skin tumour or early cervical cancer are eligible).
14. Women who are pregnant or breast feeding.
15. Stage III disease with extensive nodal disease not treatable in radical radiotherapy field.
16. Leptomeningeal disease

Eligibility Criteria for Randomisation

Following cycle 2 of induction SACT, patients must meet the following eligibility criteria for randomisation:

* No confirmed disease progression on post-cycle 2 CT scan (according to RECIST v1.1)

  * Patients with up to 5 metastases at the time of registration but less than 5 visible after induction SACT are still eligible for randomisation.
  * Patients with no visible metastases following 2 cycles of induction of SACT are eligible for randomisation. If randomised to the Investigational Arm, these patients will receive RT upon relapse of metastases (patients who experience progression with new metastases are not eligible for randomisation or for trial treatment).
  * Patients with complete response of the lung primary +/- lymph nodes following 2 cycles of induction SACT are eligible for randomisation. Patients randomised to the Investigational Arm, should receive conventional RT to the pre-SACT involved nodal stations and to any scar residuum at the primary site.
  * Patients who progress following 2 cycles of induction of SACT cannot be randomised. Only overall survival data will be collected for these patients.
* ECOG Performance Status 0-2.
* Continued suitability for trial treatment as deemed by the treating clinician.
* Continues to meet all registration eligibility criteria, as detailed in section 6.4.1 (with the exception of ECOG status).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2016-08-19 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From date of randomisation to the date of death, up to 36 months
  The trial will investigate the impact of the addition of radical conventional and stereotactic radiotherapy to standard systemic therapy on overall survival

SECONDARY OUTCOMES:
Progression Free Survival | Time from randomisation until progression or death, up to 36 months.
  The trial will investigate the impact of the addition of radical conventional and stereotactic radiotherapy to standard systemic therapy on progression free survival
Toxicity (radiotherapy related toxicity Adverse events) | From registration to up to 36 months after the first patient is randomised
  Safety analyses will be performed on all patients who received at least one dose of chemotherapy or fraction of SRT post-randomisation. Radiotherapy-related toxicity and early and late toxicity will be investigated. Adverse events will be compared between the two groups, as well as dose delays, reductions and compliance to chemotherapy and radiotherapy.
Local Tumour Control by assessment of tumours at baseline and at progression according to RECIST v1.1 | From time of randomisation to time of progression or death, up to 36 months
  The trial will investigate the impact of the addition of radical conventional and stereotactic radiotherapy to standard systemic therapy on local tumour control
Health Related Quality of Life using the EORTC-QLQ-C30 and EORTC-LC13 questionnaires | From time of registration to time of death or up to 36 months
  The health related quality of life for each treatment arm will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona McDonald, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (19):
- United Kingdom (19):
  - UCLH, London, England
  - Belfast City Hospital, Belfast
  - Queen Elizabeth Hospital, Birmingham
  - Bristol Royal Infirmary, Bristol
  - Addenbrooke's Hospital, Cambridge
  - BEATSON, Glasgow
  - Royal Surrey County Hospital, Guildford
  - St James's University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Guy's and St Thomas's Hospital, London
  - St Bart's Hospital, London
  - The Royal Marsden Hospital, London
  - Christie Hospital, Manchester
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - The James Cook University Hospital, Middlesbrough
  - Freeman Hospital, Newcastle
  - City Hospital, Nottingham
  - Weston Park Hospital, Sheffield
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Conibear J, Chia B, Ngai Y, Bates AT, Counsell N, Patel R, Eaton D, Faivre-Finn C, Fenwick J, Forster M, Hanna GG, Harden S, Mayles P, Moinuddin S, Landau D. Study protocol for the SARON trial: a multicentre, randomised controlled phase III trial comparing the addition of stereotactic ablative radiotherapy and radical radiotherapy with standard chemotherapy alone for oligometastatic non-small cell lung cancer. BMJ Open. 2018 Apr 17;8(4):e020690. doi: 10.1136/bmjopen-2017-020690. PMID 29666135